CLINICAL TRIAL: NCT01643304
Title: A Swedish Cross-sectional Study With Questionnaire to Investigate Perception of Menstrual Bleeding
Brief Title: A Swedish Questionnaire Study to Investigate the Perception of Menstrual Bleedings
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16384; NN1223SE (Other: Company Internal)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Menorrhagia
Keywords: Menorrhagia; Heavy menstrual bleeding; Uterine Hemorrhage; Menstruation Disturbancies
MeSH Terms: conditions — Menorrhagia; Uterine Hemorrhage

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Behavioral: No drug

INTERVENTIONS:
Behavioral: No drug — No drug intervention. The intervention is a questionnaire with quality of life and perception of menstrual bleedings. All subjects will complete both questionnaires.

SUMMARY:
This field based, questionnaire study will document observational data on womens perception of menstrual bleeding in a cross-section of women in Sweden. Each subject will complete the questionnaire at one occasion.

ELIGIBILITY:
Inclusion Criteria:

* All women 40-45 years available in the web-panel of SIFO
* Completion of the web-based questionnaire

Exclusion Criteria:

* None

Ages: 40 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects included in the SIFO (Swedish institute of market research) volontary subject pool.
Sampling Method: Non-Probability Sample
Enrollment: 1547 (Actual)
Dates: Start 2012-05; Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of subjectively experienced heavy menstrual bleeding assessed by questionnaire | Once at baseline

SECONDARY OUTCOMES:
Social consequences of heavy menstrual bleedings assessed by questionnaire | Once at baseline
Costs; e.g. pads, absence from work, loss of income assessed by questionnaire | Once at baseline
The treatments given for heavy menstrual bleedings, as surgery or medication assessed by questionnaire | Once at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Sweden